CLINICAL TRIAL: NCT00591045
Title: A Randomized Phase II Multicenter Controlled Study of Oxaliplatin, Calcium Folinate, and 5-Fluorouracil as Neoadjuvant Chemotherapy for Resectable Advanced Gastric Cancer
Brief Title: Study of Oxaliplatin, Calcium Folinate, and 5-Fluorouracil as Neoadjuvant Chemotherapy for Resectable Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Collaborators: Fudan University (Other); Capital Medical University (Other)
Responsible Party: Jiafu Ji, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGCCG-0701
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2007-12

CONDITIONS: Stomach Neoplasms; Gastric Cancer
Keywords: gastric adenocarcinoma; neoadjuvant chemotherapy; efficacy; safety; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The patients will undergo neoadjuvant chemotherapy with mFOLFOX and then an operation and then individualized adjuvant chemotherapy.
  Interventions: Drug: mFOLFOX
- 2 (No Intervention): No neoadjuvant chemotherapy and surgery and then adjuvant chemotherapy.

INTERVENTIONS:
Drug: mFOLFOX — oxaliplatin 100mg/m2, CF 400mg/m2, 5-FU 2400 mg/m2 46hr civ
  Arms: 1

SUMMARY:
This is a randomized phase II multicenter controlled study of oxaliplatin, calcium folinate, and 5-fluorouracil (mFOLFOX7) as neoadjuvant chemotherapy for resectable advanced gastric cancer.

Hypothesis: Neoadjuvant chemotherapy may improve 5 year overall survival compared with the control.

DETAILED DESCRIPTION:
The study hypothesis is that the 5 year survival rate will reach 35% from 25% when neoadjuvant chemotherapy is carried out. With the alpha value to be 0.05 and beta value to be 0.80 as well as 10 percent of patients' lost-of-followup, the sample size will be 263.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0-2
* Ambulatory males or females, aged 30-70 years.
* Histologically confirmed gastric adenocarcinoma, staged preoperatively AJCC/UICC stage III(T3N1,T2N2,T4N0,T3N2)and IVM0 and operable
* Life expectancy more than 3 months
* Give written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Normal hepatic, renal, and bone marrow function (GPT<2 fold of upper limit value; WBC>4000/dl, Tbil<1.5mg/dl, Cr<1.5 fold of upper limit value)

Exclusion Criteria:

* Patients can not bear surgical procedure.
* Pregnant or lactating women or women do not agree conceptive procedures.
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy except corticosteroids, for the currently treated gastric cancer.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.
* Organ allografts requiring immunosuppressive therapy.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Moderate or severe renal impairment: serum creatinine > 1.5 x upper limit of normal (ULN).
* Prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented DPD deficiency) or patients with known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Hypersensitivity to platinum compounds or any of the components of the study medications.
* Received any investigational drug or agent/procedure, i.e. participation in another trial, within 4 weeks before randomization.
* Unwilling or unable to comply with the protocol for the duration of the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
5 year overall survival | Jan 2008 to Dec 2012

SECONDARY OUTCOMES:
R0 resection rate | Jan 2008 to Dec 2012

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, M.D., Principal Investigator — Peking University
Locations (1):
- Peking University School of Oncology, Beijing, Beijing Municipality, China